CLINICAL TRIAL: NCT02005172
Title: Validation of an iPhone-based Event Recorder for Arrhythmia Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Deepika Narasimha, MD, University at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 506493-2
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Results first posted 2022-06-13 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-04

CONDITIONS: Arrhythmia, Palpitations, Lightheadedness
Keywords: arrhythmia, palpitations, lightheadedness
MeSH Terms: conditions — Arrhythmias, Cardiac; Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alivecor device and event monitor (Other): Both the Alivecor device (experimental) and the standard of care (event monitor) will be provided to all patients for the duration of the study
  Interventions: Device: Alivecor monitor and 14 day event monitor

INTERVENTIONS:
Device: Alivecor monitor and 14 day event monitor — Alivecor monitor and 14 day event monitor

SUMMARY:
In this study, we will evaluate the diagnostic yield of the new AliveCor device versus a 14 day event monitor with the use of both devices simultaneously. We will also examine by means of a questionnaire the compliance, ease of use and patient satisfaction for each device.

Hypothesis:

1. The AliveCor monitor will be non-inferior to the 14 day event monitor with respect to diagnosis of the arrhythmia responsible for a patient's symptoms.
2. The AliveCor monitor will have better compliance and acceptability compared to the 14 day event monitor, and thus there will be a greater number of days with recordings from the AliveCor monitor.

ELIGIBILITY:
Inclusion Criteria:

Patients >18 years of age with symptoms such as palpitations or pre-syncope suggestive of arrhythmias (usually occurring less frequently than once a day) with prior non-diagnostic ECGs and/or Holter monitoring.

Patients who own an iPhone 4, 4S or 5 device and demonstrate the capability of recording and uploading a test ECG recording at the office visit.

Exclusion Criteria:

1. Patients <18 years of age.
2. Patients with a myocardial infarction (MI) within the last three months, and/or known history of sustained VT/VF.
3. Patients with NYHA class IV heart failure.
4. Patients with unstable angina.
5. Patients with syncope as the presenting symptom.
6. Patients unable to or unwilling to use the device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Curtis, MD, Principal Investigator — University at Buffalo
Locations (1):
- Dent Towers, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting with palpitations (less often than daily but more frequently than several times/month) to our outpatient cardiology clinics with a nondiagnostic previous work-up (ECG and in some cases, a Holter monitor) were eligible for the study if their symptoms warranted evaluation with external loop recorders (ELRs).
Pre-assignment Details: Of the 38 patients enrolled in the study (ITT Group), 33 remained in the study (PP Group) and had monitoring data for both devices.
Groups:
- Per-Protocol (PP) Group: This group includes all patients who completed and complied with the study protocol (per-protocol [PP] sample). These patients completed monitoring with both the Alivecor device (experimental) and external loop recorder (standard of care).
Period: Overall Study
Arm/Group | Per-Protocol (PP) Group
Started | 33
ITT (This group includes the patients who met the inclusion criteria and were enrolled into the study but did not complete the study) | 38
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Thirty-eight patients were enrolled and analyzed for baseline characteristics in the intention-to-treat group. Thirty-three of those participants completed the monitoring period with the Alivecor device and the ELR. This group was identified as the pre-protocol group and the baseline characteristics for this group were separately analyzed.
Groups:
- Pre-Protocol (PP) Group: This group includes all patients who completed and complied with the study protocol (per-protocol [PP] sample).
Arm/Group | Pre-Protocol (PP) Group
Number analyzed (Participants) | 33
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 47.5 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 30
  Race: African American | 3
Educational level [Count of Participants; unit: Participants]
  High School | 5
  College | 7
  Master's | 2
  Doctorate | 1
  Not reported | 18
Symptoms [Number; unit: participants]
  Palpitations | 30
  Lightheadedness | 11
  Chest pain | 6
CAD/Previous MI [Number; unit: participants] | 4
Hypertension [Number; unit: participants] | 9
Recent ablation [Number; unit: participants] | 3
Antiarrhythmic drugs [Number; unit: participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Validation of an iPhone-based Event Recorder for Arrhythmia Detection
Description: For the primary endpoint, equivalence testing using the two one-sided test (TOST) procedure was used to compare the proportion of unpaired days in which a diagnostic recording was made with each device during the monitoring period. A difference of less than 10% between the devices on the rate of detection of arrhythmias was taken to indicate equivalence.
Time Frame: one year
Population: Intention to treat analysis
Measure: Number; unit: participants
Groups:
- Kardia Mobile (AliveCor Device): AliveCor (Kardia Mobile ) used for 14 days
- External Loop Recorder (ELR/ Event Monitor): Event monitor or ELR used for 14 days
Arm/Group | Kardia Mobile (AliveCor Device) | External Loop Recorder (ELR/ Event Monitor)
Number analyzed (Participants) | 33 | 33
participants
  Sinus tachycardia | 14 | 12
  Sinus bradycardia | 8 | 8
  Sinus arrhythmia | 5 | 2
  Sinus pause | 0 | 0
  PAC | 15 | 4
  PVC | 11 | 11
  Atrial Fibrillation | 6 | 4
  Atrial Flutter | 0 | 2
  Atrial Tachycardia | 0 | 0
  SVT | 0 | 1
  First degree AV block | 0 | 1
  Second degree AV block | 0 | 0
  Third degree AV block | 0 | 0
Statistical Analysis 1: Comparison: Kardia Mobile (AliveCor Device) vs External Loop Recorder (ELR/ Event Monitor); For the primary endpoint, equivalence testing using the two one-sided test procedure was used to compare the proportion of (unpaired) days in which a diagnostic recording was made with each device during the monitoring period. For the purpose of this study, a difference of less than 10% between devices on the rate of detection of arrhythmias was taken to indicate equivalence; Test type: Equivalence — The primary analysis used the TOST procedure for equivalence. A difference of less than 10% between devices on the proportion of diagnostic days during the monitoring period was considered to be equivalent. We hypothesized that the percentage of diagnostic days for the ELR and the KM would be 20% and 15%, respectively; Descriptive statistics (means, standard deviation (SD), percentages) were used to summarize the demographic and clinical characteristics of the patients. The total number of tracings and the percentage of tracings with arrhythmias for each device were also calculated. For the primary endpoint, equivalence testing using the two one-sided test (TOST) procedure was used to compare the proportion of (unpaired) days in which a diagnostic recording was made with each device during the monitoring period. Patients were asked to use both devices for the same duration. For the purpose of this study, a difference of less than 10% between devices on the rate of detection of arrhythmias was taken to indicate equivalence. The primary hypothesis was that the KM

ADVERSE EVENTS:
Arm/Group | Alivecor Device and Event Monitor
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No